CLINICAL TRIAL: NCT03976245
Title: Advanced Therapeutics in Rheumatoid Arthritis (RA)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Academic Medical Organization of Southwestern Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAJP0001
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Tumour Necrosis Factor; Janus kinase inhibitor
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; tofacitinib

STUDY DESIGN:
Intervention Model Description: Pragmatic, open-label, randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- etanercept (Active Comparator): etanercept 50 mg subcutaneously injected per week
  Interventions: Drug: Etanercept
- tofacitinib (Active Comparator): tofacitinib 5 mg orally daily
  Interventions: Drug: tofacitinib

INTERVENTIONS:
Drug: Etanercept — injection
  Other Names: enbrel; Brenzys
  Arms: etanercept
Drug: tofacitinib — tablet
  Other Names: Xeljanz; Jakvinus
  Arms: tofacitinib

SUMMARY:
This study will evaluate the retention rates of two advanced therapies, Tumour Necrosis Factor (TNF) and Janus kinase inhibitor (JAK) in the treatment of adults with Rheumatoid Arthritis (RA) over a two year period. It will also examine the ability to embed a clinical trial in a clinical situation using an electronic medical record (EMR).

DETAILED DESCRIPTION:
Conventional therapies for Rheumatoid Arthritis (RA) treatment include nonsteroidal anti-inflammatory drugs (NSAIDs), cyclooxygenase-2 (COX-2) selective inhibitors, corticosteroids and disease modifying anti-rheumatic drugs (DMARDs). These therapies are often partially effective.

For those patients, where conventional therapies have failed to alleviate their symptoms, Tumour Necrosis Factor (TNFis) is often prescribed to treat the pain and inflammation associated with RA. The main problem with TNFi and other advanced therapies in RA is retention. At least ¼ of patients stop treatment within a year and another ⅕ to ¼ in the second year, mostly due to secondary loss of efficacy.

Another advanced therapy, the Janus kinase inhibitor (JAK) has demonstrated similar efficacy to TNFi treatment in RA. This trial will determine if using a different class of treatment (small molecule, oral drug, JAK kinase inhibitor) will have a better retention than a TNFi (using the most commonly prescribed TNFi for RA in Canada).

ELIGIBILITY:
Inclusion Criteria:

* patients with RA who meet criteria for obtaining an advanced therapeutic through usual care
* active RA with 5 or more swollen joints
* seropositive
* presence of erosions
* failure of methotrexate and hydroxychloroquine and sulfasalazine
* failure of Leflunomide

  -> or equal to 18 years
* able to provide consent
* able to attend usual follow up visits

Exclusion Criteria:

* no contraindication to etanercept or tofacitinib
* active serious infection
* active Tuberculosis
* multiple sclerosis
* current cancer
* lymphoma ever
* previous use of an advanced therapeutic (biologic or JAK kinase inhibitor)
* less than 18 years of age
* unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Retention Rates | 24 months
  Evaluation of the proportion of patients in each arm still on the randomized treatment

SECONDARY OUTCOMES:
Mean Change in Disease Activity | 24 months
  The mean change from baseline in the Clinical Disease Activity Index in each arm of the study. The Clinical Disease Activity Index measures the number of tender or swollen joints, patient global assessment of disease activity, and provider global assessment of disease activity. Total tender joint count=0-28, total swollen joint count=0-28, patient global score=0-10, provider global score=0-10. Total range score=0-76. Higher values for all subscales, tender and swollen joints, global assessments indicate higher disease activity. Scores for subscales are combined to calculate the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Pope, MD MPH, Principal Investigator — Western University, Canada
Locations (1):
- Rheumatology Clinic, St. Joseph's Health Care, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No